CLINICAL TRIAL: NCT01632189
Title: Investigating the Effects of Varenicline on D2/3 Receptor Binding in Brain of Tobacco-smokers: a PET/[11C](+)PHNO Study
Brief Title: The Effect of Varenicline on D2/D3 Receptor Binding in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Lung Association (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Bernard Le Foll, Principal Investigator; MD, PhD, CCFP, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 040/2012
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Nicotine Dependence
Keywords: Varenicline; PET imaging; [11C]-(+)-PHNO PET; neuroimaging in smokers
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varenicline (Experimental): Varenicline will be used at the same dosage regimen as used for smoking cessation, i.e. 0.5mg once daily for days 1-3, 0.5mg twice daily for days 4-7 followed by 1mg twice daily. The total duration of Varenicline treatment will be three months.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline will be administered as prescribed: 0.5 mg for the first 3 days then 1 mg for the next 7 days and 2 mg after that. A quit date will be chosen at 11 days after starting Varenicline. Varenicline will be given for 3 months.
  Other Names: Champix

SUMMARY:
This study will evaluate effects of treatment with varenicline, a smoking cessation drug, on the dopaminergic system by using Positron Emission Tomography (PET) imaging with new radioligand, [11C]-(+)-PHNO. The investigators primary hypothesis is that chronic varenicline administration will increase dopamine (DA) receptors levels ([11C](+)PHNO) within the human brain.

DETAILED DESCRIPTION:
Subjects will undergo a pre-treatment PET and MRI scans for baseline [11C](+)PHNO measures on Day 1. Subjects will subsequently be provided an initial 2-week supply of study medications (varenicline) and directions for use. Any adverse events, compliance to medication and smoking patterns will be noted during these two weeks. Varenicline will be used at the same dosage regimen as used for smoking cessation. After subjects go through a post-treatment PET and MRI scans on Day 10, they will be instructed to set up a quit date. There will then be follow-up visits every 2 weeks for the duration of the medication phase (3 months total) and a visit at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be nicotine dependent, males and females of any ethnic origin between 21 and 45 years old.
* Meet DSM-IV criteria for nicotine dependence,
* Smoke ≥10 cigarettes/day, Baseline FTND score ≥4, CO level ≥10 and are motivated to quit within 30 days of initial intake.
* Treatment seeking smokers that are willing to use varenicline as a treatment approach for their smoking cessation attempt
* No previous use of medication for smoking cessation in previous month prior inclusion.

Exclusion Criteria:

* Pregnancy (a urine pregnancy test will be performed before each PET in women)
* Trying to become pregnant or breastfeeding;
* Have abused alcohol or other drugs of abuse (cocaine, opiates, benzodiazepines, etc) in 3 months prior to randomization.
* Presence of metal objects in the body (e.g. some artificial joints, bone pins, surgical clips, skull plate, certain part of dental braces) or implanted electronic devices (e.g. cardiac pacemaker, neurostimulator), that preclude safe MR scanning.
* Claustrophobia.
* Cardiovascular or cerebrovascular diseases.
* Major psychiatric disorders including mood, anxiety or psychotic disorders with historical evidence of suicidal or homicidal behaviour.
* History of or current neurological illnesses including seizure disorders, migraine, multiple sclerosis, movement disorders, head trauma, CVA or CNS tumor. Gross structural brain abnormalities as revealed by T1 weighted images.
* Current use or use during the previous month of medication that may affect the CNS at the time of scanning (including illicit and non-illicit psychoactive drugs).
* Learning disability, amnesia or other conditions that impede memory and attention.
* Allergy to varenicline.
* Renal insufficiency.
* Use of other smoking cessation aids

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
[11C]-(+)-PHNO DRD2/3 binding potential (BPND) | 10 days
  The effects of chronic administration of varenicline (standard dose run up protocol to 2 mg per day for 10 days) vs. baseline on [11C]-(+)-PHNO binding in human brain of tobacco smokers (12 hours abstinent).

SECONDARY OUTCOMES:
Relationship between ability to quit smoking and changes in DRD2/3 | 6 months
  Relationship between clinical ratings of abstinence and cravings and DRD2/3 normalization after 10-day course of varenicline administration.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Result] Di Ciano P, Guranda M, Lagzdins D, Tyndale RF, Gamaleddin I, Selby P, Boileau I, Le Foll B. Varenicline-Induced Elevation of Dopamine in Smokers: A Preliminary [(11)C]-(+)-PHNO PET Study. Neuropsychopharmacology. 2016 May;41(6):1513-20. doi: 10.1038/npp.2015.305. Epub 2015 Oct 7. PMID 26442600
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research